CLINICAL TRIAL: NCT02346721
Title: An Open Label Study of Sofosbuvir/GS-5816 Fixed-Dose Combination in Subjects With Chronic HCV Infection
Brief Title: Sofosbuvir/Velpatasvir Fixed-Dose Combination in Adults With Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1446; 2014-003898-42 (EudraCT Number)
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sofosbuvir; SOF/GS-5816; GS-5816; Hepatitis C; HCV; Cirrhosis; Velpatasvir
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) in participants with chronic genotype 1, 2, 4, 6 or indeterminate HCV infection who received placebo in the Gilead-sponsored study GS-US-342-1138.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
* Was administered placebo to match SOF/VEL in Gilead study GS-US-342-1138
* HCV RNA ≥ 10^4 IU/mL at screening
* Classification as treatment naive or treatment experienced
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Key Exclusion Criteria:

* Current or prior history of clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment, or compliance with the protocol; individuals currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
* Screening electrocardiogram (ECG) with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at screening
* Prior exposure to SOF or other nucleotide analogue HCV NS5B inhibitor or any HCV NS5A inhibitor
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (54):
- United States (21):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Richmond, Virginia
- Belgium (2):
  - Antwerp
  - Brussels
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Montreal, Quebec
  - Toronto
- France (11):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Toulouse
  - Villejuif
- Germany (6):
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Berlin
  - Hamburg
  - Hanover
  - München
- Hong Kong, Hong Kong
- Italy (2):
  - San Giovanni Rotondo, Foggia
  - Florence
- San Juan, Puerto Rico
- United Kingdom (6):
  - Plymouth, Devon
  - Portsmouth, Hampshire
  - Glasgow
  - London
  - Manchester
  - Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Asselah T, Shafran S, Bourgeois S, Lai CL, Cramp M, Mathurin P, et al. Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in HCV Infected Patients Previously Treated With Placebo: Results of the Deferred Treatment Study (GS-US-342-1446 Study) [Abstract SAT-279]. J Hepatology 2016;64:S827-8.
- [Derived] Asselah T, Shafran SD, Bourgeois S, Lai CL, Mathurin P, Willems B, Nguyen MH, Davis MN, Huang KC, Svarovskaia E, Osinusi A, McNally J, Brainard DM, Shaikh OS, Tran TT. Deferred treatment with a fixed-dose combination of sofosbuvir-velpatasvir for chronic hepatitis C virus genotype 1, 2, 4 and 6 infection. J Viral Hepat. 2019 Oct;26(10):1229-1232. doi: 10.1111/jvh.13159. Epub 2019 Aug 4. PMID 31216086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia Pacific. The first participant was screened on 23 February 2015. The last study visit occurred on 15 June 2016.
Pre-assignment Details: 116 participants were screened.
Groups:
- SOF/VEL 12 Weeks: Sofosbuvir/velpatasvir (SOF/VEL; Epclusa®) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily
Period: Overall Study
Arm/Group | SOF/VEL 12 Weeks
Started | 111
Completed | 107
Not Completed | 4
Not completed — Withdrew Consent | 3
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 12
  White | 85
  Asian | 11
  Native Hawaiian or Pacific Islander | 1
  Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 106
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6
  Belgium | 4
  United States | 42
  China | 1
  United Kingdom | 13
  Italy | 2
  France | 31
  Germany | 7
  Hong Kong | 3
  Puerto Rico | 2
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 36
    CT | 50
    TT | 25
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.55)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 30
  ≥ 800,000 IU/mL | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set (FAS) included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL 12 Weeks: SOF/VEL 400/100 mg FDC tablet orally once daily
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
percentage of participants | 97.3 [92.3 to 99.4]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
percentage of participants | 0.9

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
percentage of participants
  SVR4 | 98.2 [93.6 to 99.8]
  SVR24 | 97.3 [92.3 to 99.4]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL 12 Weeks: SOF/VEL 400/100 mg fixed-dose combination (FDC) tablet orally once daily
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
percentage of participants
  Week 1 | 18.0 [11.4 to 26.4]
  Week 2 | 55.0 [45.2 to 64.4]
  Week 4 | 94.6 [88.6 to 98.0]
  Week 6 | 99.1 [95.1 to 100.0]
  Week 8 | 100.0 [96.7 to 100.0]
  Week 10 | 100.0 [96.7 to 100.0]
  Week 12: number analyzed (Participants) | 110
  Week 12 | 100.0 [96.7 to 100.0]

5. Secondary Outcome: HCV RNA Change From Baseline
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 110
  Change at Week 1 | -4.23 (0.592)
  Change at Week 2 | -4.79 (0.627)
  Change at Week 4 | -5.10 (0.546)
  Change at Week 6 | -5.11 (0.552)
  Change at Week 8 | -5.11 (0.554)
  Change at Week 10 | -5.11 (0.554)
  Change at Week 12: number analyzed (Participants) | 110
  Change at Week 12 | -5.11 (0.556)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 111
percentage of participants | 0.9

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL 12 Weeks
Serious Adverse Events (participants affected / at risk) | 5/111
Other Adverse Events (participants affected / at risk) | 46/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (N=111)
Cellulitis (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (N=111)
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 18
Headache (Nervous system disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years